CLINICAL TRIAL: NCT07384442
Title: Effects of Targeted Temporal Interference Stimulation of Cerebellar Nuclei on Tremor and Gait Disturbance in Parkinson's Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YangPan (Other)
Responsible Party: Sponsor-Investigator, YangPan, Zhongnan Hospital, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2026022
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease; Movement Disorders
Keywords: Parkinson's Disease; Cerebellar Nuclei; Movement Disorders; Tremor; Gait; Temporal Interference Stimulation
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Comparator (Sham Comparator): Sham stimulation targeting the cerebellar nuclei
  Interventions: Device: Sham Temporal Interference Stimulation
- Active Comparator (Active Comparator): Real TIS targeting the cerebellar nuclei
  Interventions: Device: Real Temporal Interference Stimulation

INTERVENTIONS:
Device: Sham Temporal Interference Stimulation — Patients will be randomly allocated into this group, and they will receive sham TIS-targeted stimulation of cerebellar nuclei, stimulating both sides of the cerebellum daily for 20 minutes each side. Start with the left side, immediately followed by the right side upon completion, totaling 40 minutes of stimulation. Continue this cycle for 5 days, followed by 2 days of rest, then repeat for another 5 days, repeating this process continuously for 19 days.The TIS frequency was set to 0 Hz to prevent the generation of envelope currents.
  Arms: Sham Comparator
Device: Real Temporal Interference Stimulation — Patients will be randomly allocated into this group, and they will receive real stimulation.TIS-targeted stimulation of cerebellar nuclei, stimulating both sides of the cerebellum daily for 20 minutes each side. Start with the left side, immediately followed by the right side upon completion, totaling 40 minutes of stimulation. Continue this cycle for 5 days, followed by 2 days of rest, then repeat for another 5 days, repeating this process continuously for 19 days. The TIS was set at a frequency of 100 Hz; The stimulus frequency difference was fixed for each subject, while the stimulus current was adjusted based on individual tolerance and clinical needs.
  Arms: Active Comparator

SUMMARY:
The goal of this clinical trial is to explore the effects of cerebellar nuclei TIS stimulation on improving tremor and gait disorders in PD patients. Through randomized double-blind grouping, the differences in efficacy between TIS intervention and sham stimulation intervention for tremor and gait disorders in PD patients will be compared.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder with an extremely high global incidence rate and is also one of the most common movement disorders. The core motor symptoms of this disease are particularly complex, encompassing various specific clinical features, including bradykinesia, resting tremor, muscle rigidity, and postural and gait disturbances. The progressive worsening of these symptoms is closely associated with the gradual loss of dopaminergic neurons in the substantia nigra-striatal pathway of the brain, which directly leads to significant impairment of motor control function. In recent years, with the continuous advancement of neuroimaging techniques and electrophysiological research methods, scientists have gradually revealed the critical role of the cerebellum in the pathophysiological mechanisms of Parkinson's disease. Studies have shown that the cerebellum is not only a key node in the motor control network but also deeply involved in the pathogenesis of PD tremor through the thalamocortical circuit. Additionally, the cerebellum plays an indispensable role in regulating gait stability through functional connections with the basal ganglia and cerebral cortex. Based on the dual role of the cerebellum in the pathophysiological processes of Parkinson's disease, this study plans to employ an innovative technical approach-targeted temporal interference stimulation (TIS) of cerebellar nuclei-to precisely modulate the activity of cerebellar neural circuits in a non-invasive manner. The cerebellar nuclei are located deep within the white matter of the cerebellum and can be further subdivided into the dentate nucleus, intercalated nucleus, and vermis, which exhibit distinct differences from the cerebellar cortex. As the core output hub of the entire cerebellum, all signals originating from the cerebellar cortex ultimately converge here before being projected to the cerebral cortex, brainstem, and spinal cord, regulating motor coordination, gait, balance, muscle tone, and tremors. Transcranial induction stimulation (TIS) non-invasively modulates the intact cerebellar nuclei, enabling direct regulation of cerebellar function, which is more efficient compared to modulating the cerebellar cortex.

The objective of this intervention approach is to validate its efficacy in improving tremor and gait disorders in patients with Parkinson's disease (PD), thereby providing a novel neuromodulatory strategy for the clinical treatment of motor symptoms in PD and further expanding our understanding and application scope of therapeutic approaches for this disorder.

To explore the effect of TIS targeting cerebellar nuclei on tremor and gait disorders in PD patients. Participants will be assigned to group active TIS/sham TIS by using the method of generating random numbers and receive:

1. Unified Parkinson Disease Rating Scale (UPDRS) before and after the treatment course.
2. Zhenluo Gait Device evaluation.
3. Electromyography tremor assessment Researchers will compare the data collected from UPDRS, Zhenluo Gait Device analysis, and electromyography tremor assessment rating between the active TIS group and sham controls before and after the treatment to see if there are meliorating effects of TIS on Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 50 years or older;
* 2.Confirmed diagnosis of idiopathic Parkinson's disease (IPD) according to the 2015 MDS diagnostic criteria, with tremor and gait disturbance;
* 3.Disease duration ≥2 years after diagnosis, stable condition, and ability to cooperate with study assessment and intervention;
* 4.Stable medication dosage for at least 4 weeks prior to the trial;
* 5.Good response to Levodopa therapy;
* 6.Capable of independent walking (without assistive devices) for at least 5 minutes and able to complete gait testing independently.
* 7.Signed informed consent form, with the participant or their legal guardian able to understand and willing to participate in this study.

Exclusion Criteria:

* 1.History or confirmed diagnosis of severe mental disorders, such as depression, anxiety disorders, schizophrenia spectrum disorders, and bipolar disorder;
* 2.The subject has clinically defined neurological conditions (assessed through self-report), including but not limited to: any disease potentially associated with increased intracranial pressure, space-occupying lesions, stroke history, transient ischemic attack (TIA) within the past two years, cerebral aneurysm, dementia, multiple sclerosis;
* 3.Severe cognitive impairment, Mini-Mental State Examination (MMSE) score <22, or inability to independently complete questionnaires;
* 4.Inability to read or understand Chinese;
* 5.Use of other neuromodulatory therapies within the past 3 months;
* 6.Presence of musculoskeletal or orthopedic conditions (e.g., severe arthritis, recent fractures) that significantly interfere with gait or balance;
* 7.Presence of metal implants (e.g., Deep Brain Stimulation, cardiac pacemakers) or contraindications for MRI/TIS;
* 8.Current use of medications that affect dopamine levels (e.g., antipsychotics);
* 9.Severe cardiovascular disease or other unstable medical conditions that preclude physical exertion or study participation;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of electromyographic tremor index | Baseline, at the end of the 19-day post-treatment, 30-day follow up.
  The values of the tremor amplitude (oscillatory displacement) will be collected from each participant to measure the intensity of the tremor with values ranging from 0 mm (absence of tremor) to the peak amplitude (maximum intensity). The higher values mean a worse motor stability.
Changes of Zhenluo Gait Device evaluation | Baseline, at the end of the 19-day post-treatment, 30-day follow up.
  The parameters of the Zhenluo Gait Device evaluation (spatiotemporal gait analysis) will be collected from each participant to measure the stability and quality of walking patterns with values ranging from pathological (abnormal deviation) to physiological (normal gait). The greater deviation from normative data means a worse gait performance.

SECONDARY OUTCOMES:
Changes in the scores of the UPDRS | Baseline, at the end of the 19-day post-treatment, 30-day follow up.
  The UPDRS (total) score will be collected from each participant to measure the overall severity of Parkinson's disease, with scores ranging from 0 (minimum) to 199 (maximum). The higher scores mean a worse outcome.